CLINICAL TRIAL: NCT03857516
Title: Multipolar Left Ventricular Electrode Instability Trial
Acronym: MOVE IT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-022
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Pacemaker Electrode Lead Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recipients of cardiac resynchronization therapy: Consecutive patients with de novo implantation of a cardiac resynchronization defibrillator or pacemaker.
  Interventions: Device: Multipolar left ventricular lead implantation

INTERVENTIONS:
Device: Multipolar left ventricular lead implantation — Multipolar left ventricular lead implantation with measurements of pacing thresholds in varrious pacing configurations.

SUMMARY:
Characterization of pacing thresholds in available pacing vectors of quadripolar leads used for cardiac resynchronization therapy in a short term follow-up.

DETAILED DESCRIPTION:
Multipolar left ventricular leads are increasingly used in cardiac resynchronization therapy. Lead dislodgment requiring re-intervention is rare. However, data on minor lead movements which may affect pacing capabilities and application of new pacing algorithms is scarce. Aim of the study is to characterize pacing thresholds of each of the implanted electrodes on quadripolar leads in a short term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* De novo implantation of left ventricular multipolar leads.

Exclusion Criteria:

* Cardiogenic shock
* Device infection
* Revision for previously dislodged left ventricular lead
* Age below 18 years
* Pregnancy
* Patients under tutelage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving cardiac resynchronization therapy according to guidelines with the implantation of a multipolar left ventricular lead.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Microdislodgement of leads | 3 months
  Change of pacing threshold

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches herzzentrum Muenchen, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No